CLINICAL TRIAL: NCT07356661
Title: Randomized Double-blind Placebo-controlled Study of the Evaluation of the Efficacy of Neurofeedback Technique Based on EEG Desynchronization in Pharmaco-resistant Epilepsy
Brief Title: Evaluation of the Efficacy of Neurofeedback Technique Based on EEG Desynchronization in Epileptic Patients
Acronym: EPIFEED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCAPHM22_0313; ID-RCB 2025-A00981-48 (Other: ANSM)
Record Dates: First submitted 2025-09-27; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Epilepsy; Drug Resistant Epilepsy
Keywords: epilepsy; neurofeedback; connectivity
MeSH Terms: conditions — Epilepsy; Drug Resistant Epilepsy | interventions — Neurofeedback; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NFB-FC (Experimental)
  Interventions: Procedure: Neurofeedback
- Sham-NFB (Placebo Comparator)
  Interventions: Procedure: Sham-NFB

INTERVENTIONS:
Procedure: Neurofeedback — The intervention will consist of 12 training sessions at the hospital conducted with the assistance of a nurse. Each session will last approximately 40 minutes, with two resting EEG phases at the beginning and end of the session. The NFB procedure will consist of 6 training blocks of 75 seconds separated by 15-second rest blocks and 15-second baseline blocks. The patient will then be required to practice what they have learned at home.
  Other Names: Questionnaires
  Arms: NFB-FC
Procedure: Sham-NFB — The intervention will consist of 12 training sessions at the hospital conducted with the assistance of a nurse. Each session will last approximately 40 minutes, with two resting EEG phases at the beginning and end of the session. The NFB procedure will consist of 6 training blocks of 75 seconds separated by 15-second rest blocks and 15-second baseline blocks. The patient will then be required to practice what they have learned at home.
  Arms: Sham-NFB

SUMMARY:
A large proportion of patients (approximately 30%) with drug-resistant epilepsy are not eligible for surgical treatment. The alternatives that can be offered to reduce the frequency of seizures are neuromodulation (vagus nerve stimulation (VNS), deep brain stimulation (DBS), or transcranial direct current stimulation (tDCS)). Most of these alternatives require invasive procedures and therefore carry risks.

Neurofeedback (NFB) is a potential adjunctive treatment that allows patients to self-modulate brain activity and thus reduce seizure frequency in a non-invasive manner.

This technique involves measuring neurophysiological activity using a technical interface to extract a parameter of interest, which is presented in real time to the participant, who has been trained and has learned how to modify it.

NFB is of interest in various neurological and psychiatric diseases and can lead to improvement in mood disorders, which are frequently associated with epilepsy. Previous NFB methods in epilepsy aimed to modulate sensorimotor rhythms or slow cortical potentials. The investigators propose an innovative EEG-NFB paradigm based on real-time estimation of EEG functional connectivity (FC) measured on the scalp EEG (NFC-FC).

This paradigm was developed based on previous studies demonstrating increased functional brain connectivity during the interictal period and decreased synchrony induced by VNS and transcranial electrical stimulation as a possible anti-epileptic mechanism.

This study consists of a randomized, double-blind comparison between NFB-FC and sham-NFB (control). The effect of this functional connectivity-based NeuroFeedBack (NFB-FC) will be evaluated on the number of seizures before and after treatment, as well as on their severity and on criteria related to quality of life.

In this study, two healthy volunteers will be recruited in order to generate the sham sessions.

ELIGIBILITY:
For patients :

Inclusion Criteria:

* Male or female patient between 18 and 65 years old
* Patient suffering from focal or multifocal drug-resistant epilepsy
* Patient having a number of seizures: at least 3 / month during the baseline
* Patient's IQ, which in the investigator's opinion will enable questionnaires and neuropsychological assessments to be carried out;
* Patient having stable medications for epilepsy 4 weeks before the baseline (except rescue treatment);
* Patient able to understand, speak and write in French;
* Patient willing to participate, and gave written consent to the study after receiving clear information
* Patient beneficiary or affiliated to a health insurance plan

Exclusion Criteria:

* - Difficulty reading or understanding the French language or inability to understand information about the study
* Generalized epilepsy
* Major visual impairment incompatible with the realization of neurofeedback, based on investigator's opinion.
* Patient currently having psychogenic non-epileptic seizures
* Any condition that makes the study subject, in the opinion of the investigator, unsuitable for the study including presence of any disease, abnormality, medical or physical condition that, in the opinion of the investigator, may adversely impact, compromise, interfere, limit, affect or reduce the safety of the subject, the integrity of the data ; Person protected by articles L1121-5, L1121-6 of Public Health Code (pregnant or breastfeeding woman, deprived of liberty by judicial decision, situations of social fragility, adults unable or unable to express their consent, person under judicial safeguard (article L1122-2)).

For healthy volunteers :

Inclusion criteria :

* Male or female of over 18 years of age
* IQ compatible with the realization of the study
* Patient able to understand, speak and write in French;
* Patient willing to participate, and gave written consent to the study after receiving clear information
* Subject beneficiary or affiliated to a health insurance plan

Exclusion criteria :

* Subject presenting any neurological or psychiatric illnesses.
* Subject having major visual impairment incompatible with the realization of neurofeedback, based on investigator's opinion.

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of NFB-FC training on seizure frequency | 3 months after the end of the training vs 3 months before training
  Comparison to the NFB-sham training calculated in the pre-training period of reference

SECONDARY OUTCOMES:
To compare between groups the psychiatric impact (depression and anxiety) | 3-months after the end of the training
  Changes between groups of psychiatric comorbidities, specifically depression: score of the NDDI-E (Neurological Disorders Depression Inventory for Epilepsy, 6 to 24, 24 meaning bad outcome) and anxiety: Score of GAD-7 (between 0 and 21, 21 meaning bad outcome)
To compare between groups the cognitive impact | One year after inclusion
  EpiTrack evaluation
To compare between groups the quality of life | 3-months after the end of the training to the pre-training period
  QOLIE scale (Quality of Life in Epilepsy Inventory-Form 31, 0 to 100, 100 being the best outcome)
To compare between groups the number of responders | 3-months after the end of the training
  Patients showing a reduction in seizure frequency>50%
To compare between groups the number of seizure-free patients | 3-months after the end of the training
  Number of patients free of seizures
To compare between groups the change in seizure severity | 3-months after the end of the training
  Score of seizure severity (NHS3, National Hospital Seizure Severity Scale, 1 to 27, 27 being the worst outcome)
The impact of transfer skills | 6 weeks of applied learned strategies
  Use of the diary of seizures the Score of seizure severity
To assess, in the whole sample and per group (sham, active), correlations between FC changes and clinical outcomes | At the end of the training and at 3 months after the end of the training
  Comparison of coherence values between the first recording (before the first session) and the last recording (after the last session) between responders and non-responders
To assess, in the whole sample and per group (sham, active), correlations between FC changes and clinical outcomes | At 3 months after the end of the training
  Comparison of coherence values between the first recording (before the first session) and the last recording (after the last session) between responders and non-responders
To assess, in the whole sample and per group (sham, active), neurophysiological correlations, psychosocial factors and mental strategies and clinical outcomes. | At 3 months after the end of the training
  Score of mindfulness (FMI-fr); the Score of subjective cognitive state during NFB (NExT-Q), the Score of expectation and locus of control (Exp-LoC-Q),the Score of metacognition (Metacogn-IQ) and clinical outcome (seizure frequency, severity of seizures).
To assess, in the whole sample and per group (sham, active), neurophysiological correlations, psychosocial factors and mental strategies and clinical outcomes. | After each training sessions
  Score of mindfulness (FMI-fr); the Score of subjective cognitive state during NFB (NExT-Q), the Score of expectation and locus of control (Exp-LoC-Q),the Score of metacognition (Metacogn-IQ) and clinical outcome (seizure frequency, severity of seizures).

IPD SHARING:
Plan to Share IPD: No